CLINICAL TRIAL: NCT00958633
Title: Mood Stabilizer Plus Antidepressant Versus Mood Stabilizer Plus Placebo in the Maintenance Treatment of Bipolar Disorder
Brief Title: Mood Stabilizer (MS)+ Antidepressant vs MS + Placebo in Maintenance of Bipolar Disorder.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was stopped before the planned sample size was reached owing to the Covid-19 pandemic and expiration of funding.
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry); Lundbeck Canada Inc. (Industry); Lupin Limited (Industry)
Responsible Party: Principal Investigator, Lakshmi N Yatham, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H09-01017
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I disorder; Depression; Antidepressant
MeSH Terms: conditions — Depression | interventions — Escitalopram; Dexetimide; Bupropion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 8 week arm (Active Comparator): During the double-blind phase, all patients will continue treatment with their anti-manic medication(s)and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 1 patients randomized to the "8 week arm" will discontinue antidepressant treatment after 8 weeks, as recommended in current clinical practice guidelines. The antidepressant will be tapered in a double-blind manner beginning at 6 weeks, and will be substituted with placebo by 8 weeks.
  Escitalopram 10 - 30 mg or Bupropion XL 150 - 450 mg
  Interventions: Drug: Escitalopram; Drug: Bupropion XL
- 52 week arm (Active Comparator): During the double-blind phase, all patients will continue treatment with their anti-manic medication(s) and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 2 patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.
  Escitalopram 10 - 30 mg or Bupropion XL 150 - 450 mg
  Interventions: Drug: Escitalopram; Drug: Bupropion XL

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be prescribed in the dose range 10-30 mg daily.
  In patients randomized to the "8-week group:
  * escitalopram will be tapered, discontinued, and replaced with placebo over a period of 2 weeks, beginning at the week 6 study visit. The dose of escitalopram (or matching placebo) may be decreased in 10 mg increments only in the case of intolerable side effects. The dose must remain within the protocol-defined range of 10-30 mg daily at all time points.
  Patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.
  Other Names: Lexapro/Cipralex
Drug: Bupropion XL — Bupropion XL will be prescribed in the dosage range 150-450 mg daily.
  In patients randomized to the "8-week group:
  * bupropion XL will be tapered, discontinued, and replaced with placebo over a period of 2 weeks, beginning at the week 6 study visit. The dose of bupropion XL (or matching placebo) may be decreased in 150 mg increments only in the case of intolerable side effects. The dose must remain within the protocol-defined range of 150-450 mg daily at all time points.
  Patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.
  Other Names: Wellbutrin

SUMMARY:
Patients with bipolar I disorder (BD) experience depression 3 times more frequently than mania, and antidepressants are prescribed as adjuncts to mood stabilizers in up to 70% of patients. However, no placebo-controlled trials have assessed the efficacy or safety of modern antidepressants in combination with mood stabilizers in the maintenance treatment of BD. The investigators propose a multicentre, randomized, double-blind clinical trial comparing mood stabilizer plus antidepressant (escitalopram or bupropion XL) to mood stabilizer plus placebo in the maintenance treatment of BD.

The investigators hypothesize that in clinically representative patients with bipolar disorder, who respond to acute treatment with a newer antidepressant medication in conjunction with a mood stabilizing medication, continuing the antidepressant for 12 months will reduce the risk of relapse into any mood episode, including depression, mania, and hypomania, compared to stopping the antidepressant after 8 weeks.

DETAILED DESCRIPTION:
Study Design:

The investigators propose a multicentre, randomized, double-blind, placebo-controlled trial in patients with BD who are currently experiencing a depressive episode. The trial will consist of two phases: an open-label acute treatment phase, and a double-blind maintenance treatment phase.

OPEN-LABEL ACUTE TREATMENT PHASE

Experimental Design Patients with BD depression who are receiving treatment with antimanic medication(s), defined as: 1) a mood stabilizer (lithium or divalproex ), 2) a second-generation antipsychotic (SGA) (risperidone, olanzapine, quetiapine, aripiprazole, or ziprasidone), or 3) combination anti-manic therapy (two mood stabilizers; or a mood stabilizer plus an SGA (the SGA asenapine will also be permitted if prescribed with a mood stabilizer); or a mood stabilizer or SGA plus lamotrigine), will have open-label escitalopram 10-30 mg/day or bupropion XL 150-450 mg/day added to their medication(s) for up to 16 weeks.Patients who complete at least 4 weeks of treatment and achieve remission from their index depression which is maintained for ≥ 2 weeks will be eligible to enter the double-blind study phase. The duration of treatment in the open-label phase will be 4-16 weeks, depending on the time required to achieve remission.

DOUBLE-BLIND MAINTENANCE TREATMENT PHASE

Patients who are in remission from their index depression for ≥ 2 weeks and ≤ 8 weeks are eligible to take part in the double-blind maintenance phase. There are two routes to enter the double-blind phase:

* following completion of the open-label phase, or
* following a period of clinical treatment, not exceeding 16 weeks, with the same medications used in the open-label phase. Patients who respond to clinical treatment with carbamazepine plus an antidepressant may also enter the double-blind phase.

Experimental Design

During the double-blind phase, all patients will continue treatment with their anti-manic medication(s) and will be randomized to one of two treatment arms for up to 52 weeks:

* Patients randomized to the "8 week arm" will discontinue antidepressant treatment after 8 weeks, as recommended in current clinical practice guidelines..
* Patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

OPEN-LABEL ACUTE TREATMENT PHASE

1. Diagnosed with BD, current episode depressed, with a MADRS score ≥ 20 at both the screening and baseline assessments
2. The duration of the current depressive episode is ≥ 2 weeks but ≤ 52 weeks
3. Taking or initiating treatment with an anti-manic medication at a therapeutic dose. Anti-manic medications and therapeutic doses are: lithium, serum level 0.6-1.4 mEq/L; divalproex, serum level 350-700 mM; risperidone 1-6 mg/day; olanzapine 5-30 mg/day; quetiapine IR or XR 300-900 mg/day; aripiprazole 10-30 mg/day; and ziprasidone 80-160 mg/day. Combinations of these medications as outlined above, or the combination of any of them with lamotrigine 100-400 mg daily, or the combination of a mood stabilizer plus asenapine 5-20 mg/day, are also permitted.
4. If taking any other psychoactive medication (other than lorazepam ≤ 4 mg/day or equivalent), is agreeable to tapering and discontinuing it over a period of ≤ 4 weeks
5. If female and of childbearing potential, is using an adequate method of contraception.
6. Aged 18-70 years, inclusive
7. Fluent in English and capable of providing informed consent

DOUBLE-BLIND MAINTENANCE TREATMENT PHASE

• Patients meeting all of the following criteria will be eligible to be included in the double-blind study phase:

1. Taking escitalopram 10-30 mg/day or bupropion XL 150-450 mg/day, in addition to their anti-manic medication.
2. Has adequately tolerated the combination of antidepressant plus mood stabilizer, and is currently in remission for ≥ 2 weeks and ≤ 8 weeks
3. If female and of childbearing potential, is using an adequate method of contraception

Exclusion Criteria:

OPEN-LABEL ACUTE TREATMENT PHASE

1. Has a history of rapid cycling, defined as ≥ 4 mood episodes in the preceding 12 months
2. Has current manic, hypomanic, or subsyndromal hypomanic symptoms, defined as a Young Mania Rating Scale (YMRS) score ≥ 8 at the screening or baseline visits
3. Has previously been refractory to treatment with both escitalopram and bupropion XL, or has been unable to tolerate both medications due to intolerable side effects or an allergic reaction
4. Is taking monoamine oxidase inhibitors, such as phenelzine or tranylcypromine
5. Escitalopram is contraindicated in patients taking pimozide or ziprasidone. Patients on pimozide or ziprasidone can participate in the study and will be prescribed bupropion XL
6. Bupropion XL is contraindicated in patients taking other preparations containing bupropion, in patients with active eating disorders, including anorexia nervosa and bulimia nervosa; and in patients with seizure disorders. Patients with any of these can still participate in the study and will be prescribed Escitalopram
7. Has active substance dependence, other than caffeine or nicotine dependence, in the preceding 3 months. Otherwise, patients with comorbid substance abuse or other comorbid psychiatric illnesses will be eligible to participate in the study
8. Is at high risk for suicide, as defined by a score of ≥ 4 on the suicide item of the MADRS, or in the opinion of the investigator
9. Has an unstable medical illness, as defined by a change in medication or other treatment in the past 4 weeks, or in the opinion of the investigator
10. Has significant abnormalities on an electrocardiogram
11. Is pregnant or lactating

DOUBLE-BLIND MAINTENANCE TREATMENT PHASE

1. Has a history of rapid cycling, defined as ≥ 4 mood episodes in the preceding 12 months
2. Has current manic, hypomanic, or subsyndromal hypomanic symptoms, defined as a YMRS score ≥ 8 at the screening or baseline visits
3. Has active substance dependence, other than caffeine or nicotine dependence, in the preceding 3 months. Otherwise, patients with comorbid substance abuse or other comorbid psychiatric illnesses will be eligible to participate in the study
4. Is at high risk for suicide, as defined by a score of ≥ 4 on the suicide item of the MADRS, or in the opinion of the investigator
5. Has an unstable medical illness, as defined by a change in medication or other treatment in the past 4 weeks, or in the opinion of the investigator.
6. Has significant abnormalities on an electrocardiogram
7. Is pregnant or lactating
8. Has experienced an episode of mania, hypomania, or a mixed episode during antidepressant treatment of the acute depression, defined as a YMRS score of ≥ 16 at any open-label study visit, or in the opinion of the study psychiatrist

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2010-11; Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Yatham, Dr., Principal Investigator — University of British Columbia; B. Frey, Dr., Study Director — St. Joseph's Healthcare, Hamilton, Ont.; S. Beaulieu, Dr., Study Director — Douglas Mental Health University Institute, Montreal, Quebec; A. Daigneault, Dr., Study Director — Douglas Mental Health University Institute, Montreal, Quebec; A. Ravindran, Dr., Study Director — Centre for Addictions and Mental Health, Toronto, Ont.; A. Schaffer, Dr., Study Director — Sunnybrook Health Sciences Centre, Toronto, Ont.; R. Milev, Dr., Study Director — Queen's University, Kingston, Ontario; P. Cervantes, Dr., Study Director — McGill University Health Centre, Montreal, Que; T. H. Ha, Dr., Study Director — Seoul National University Bundang Hospital; Y. M. Ahn, Dr., Study Director — Seoul National University Hospital; Y. H. Joo, Dr., Study Director — Asan Medical Centre, Korea; S. Won, Dr., Study Director — Kyungpook National University Hospital, Korea; J. Y. Reddy, Dr., Study Director — National Institute of Mental Health and Neuro sciences, Bangalore, India; P.S. Sharma, Dr., Study Director — Kasturba Medical College Manipal, India; M.S. Reddy, Dr., Study Director — Asha Hospital, Hyderabad, India; A.V. Mysore, Dr., Study Director — St. John's hospital, Bangalore, India
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yatham LN, Arumugham SS, Kesavan M, Ramachandran K, Murthy NS, Saraf G, Ouyang Y, Bond DJ, Schaffer A, Ravindran A, Ravindran N, Frey BN, Daigneault A, Beaulieu S, Lam RW, Kondapuram N, Reddy MS, Bhandary RP, Ashok MV, Ha K, Ahn YM, Milev R, Wong H, Reddy YCJ; BEAM-BD Trial Group. Duration of Adjunctive Antidepressant Maintenance in Bipolar I Depression. N Engl J Med. 2023 Aug 3;389(5):430-440. doi: 10.1056/NEJMoa2300184. PMID 37530824

RESULTS

PARTICIPANT FLOW:
Groups:
- 8 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s)and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 1 patients randomized to the "8 week arm" will discontinue antidepressant treatment after 8 weeks, as recommended in current clinical practice guidelines. The antidepressant will be tapered in a double-blind manner beginning at 6 weeks, and will be substituted with placebo by 8 weeks.
  Escitalopram 10 - 30 mg daily or Bupropion XL 150 - 450 mg daily
  * In patients randomized to the "8-week group", escitalopram/bupropion will be tapered, discontinued, and replaced with placebo over a period of 2 weeks, beginning at the week 6 study visit.
- Open-Label Phase (up to 16 Weeks): Patients with BD depression who are receiving treatment with antimanic medication(s) will have open-label escitalopram 10-30 mg/day or bupropion XL 150-450 mg/day added to their medication(s) for up to 16 weeks.
Period: Open-Label (up to 16 Weeks)
Arm/Group | 8 Week Arm | 52 Week Arm | Open-Label Phase (up to 16 Weeks)
Started | 0 | 0 | 209
Completed | 0 | 0 | 150
Not Completed | 0 | 0 | 59
Not completed — Lost to Follow-up | 0 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 18
Not completed — Worsening of symptoms | 0 | 0 | 13
Not completed — Lack of Efficacy | 0 | 0 | 8
Not completed — Non-adherence | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 4
Period: Double-Blind Phase (up to 52 Weeks)
Arm/Group | 8 Week Arm | 52 Week Arm | Open-Label Phase (up to 16 Weeks)
Started (28 participants entered directly into the double-blind phase and 150 entered from the OL phase. 178 participants were randomized in the double-blind phase of which 1 was excluded due to missing baseline and follow-up data) | 88 | 90 | 0
Completed | 87 | 90 | 0
Not Completed | 1 | 0 | 0
Not completed — Excluded due to missing baseline and follow-up data. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Some participants who took part in the Open Label Phase were then included in the Double Blind portion of the study therefore certain participants are represented more than once in the Total Arm/Group.
  Final analysis 8 week arm - 87 participants. Excluded one participant due to missing baseline and follow-up data.
  52 week arm - 90 participants.
Groups:
- Double-blind 8 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s)and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 1 patients randomized to the "8 week arm" will discontinue antidepressant treatment after 8 weeks, as recommended in current clinical practice guidelines. The antidepressant will be tapered in a double-blind manner beginning at 6 weeks, and will be substituted with placebo by 8 weeks.
  Escitalopram 10 - 30 mg daily or Bupropion XL 150 - 450 mg daily
- Double-blind 52 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s) and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 2 patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.
  Escitalopram 10 - 30 mg daily or Bupropion XL 150 - 450 mg daily
- Open-Label Phase (4-16 Weeks): Patients with BD depression who are receiving treatment with antimanic medication(s) will have open-label escitalopram 10-30 mg/day or bupropion XL 150-450 mg/day added to their medication(s) for up to 16 weeks.Patients who complete at least 4 weeks of treatment and achieve remission from their index depression which is maintained for ≥ 2 weeks will be eligible to enter the double-blind study phase. The duration of treatment in the open-label phase will be 4-16 weeks, depending on the time required to achieve remission.
- Total: Total of all reporting groups
Arm/Group | Double-blind 8 Week Arm | Double-blind 52 Week Arm | Open-Label Phase (4-16 Weeks) | Total
Number analyzed (Participants) | 87 | 90 | 206 | 383
Age, Categorical [Count of Participants; unit: Participants] — Population: Some participants who took part in the Open Label Phase were then included in the Double Blind portion of the study.
  Participants
    Double-blind 8 week and 52 week arm: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-blind 8 week and 52 week arm: <=18 years | 0 | 0 | 0 | 0
    Double-blind 8 week and 52 week arm: Between 18 and 65 years | 87 | 90 | 0 | 177
    Double-blind 8 week and 52 week arm: >=65 years | 0 | 0 | 0 | 0
    Open-Label 4-16 week arm: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label 4-16 week arm: <=18 years | 0 | 0 | 0 | 0
    Open-Label 4-16 week arm: Between 18 and 65 years | 0 | 0 | 206 | 206
    Open-Label 4-16 week arm: >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are being reported separately for the Open-label and Double-Blind arms.
  years
    Double-Blind Phase: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-Blind Phase | 42.9 (11.1) | 39.3 (11.3) |  | 41.1 (11.3)
    Open-Label Phase: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label Phase |  |  | 40.1 (10.9) | 40.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are being reported separately for the Open-label and Double-Blind arms.
  Participants
    Double-blind 8 week arm: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-blind 8 week arm: Female | 48 | 44 | 0 | 92
    Double-blind 8 week arm: Male | 39 | 46 | 0 | 85
    Open-Label Phase: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label Phase: Female | 0 | 0 | 107 | 107
    Open-Label Phase: Male | 0 | 0 | 99 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data are being reported separately for the Open-label and Double-Blind arms.
  Participants
    Double-Blind Phase: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-Blind Phase: Asian | 76 | 78 |  | 154
    Double-Blind Phase: Black | 1 | 0 |  | 1
    Double-Blind Phase: White | 10 | 11 |  | 21
    Double-Blind Phase: Other | 0 | 1 |  | 1
    Open-Label Phase: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label Phase: Asian |  |  | 176 | 176
    Open-Label Phase: Black |  |  | 1 | 1
    Open-Label Phase: White |  |  | 28 | 28
    Open-Label Phase: Other |  |  | 1 | 1
Montgomery Asberg Depression Rating Scale Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a scale measuring depression severity. The scale ranges from a minimum value of 0 to a maximum value 60. A higher score means a worse outcome. Population: Data are being reported separately for the Open-label and Double-Blind arms.
  units on a scale
    Double-Blind Phase: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-Blind Phase | 3.2 (2.0) | 3.1 (2.5) |  | 3.2 (2.3)
    Open-Label Phase: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label Phase |  |  | 26.6 (4.9) | 26.6 (4.9)
Drug Combination - No. [Count of Participants; unit: Participants] — Population: Data are being reported separately for the Open-label and Double-Blind arms.
  Participants
    Double-Blind Phase: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-Blind Phase: Bupropion XL plus Mood Stabilizer | 17 | 16 |  | 33
    Double-Blind Phase: Bupropion XL plus Mood Stabilizer plus SGA | 14 | 16 |  | 30
    Double-Blind Phase: Bupropion XL plus SGA | 1 | 3 |  | 4
    Double-Blind Phase: Escitalopram plus Mood Stabilizer | 24 | 24 |  | 48
    Double-Blind Phase: Escitalopram plus Mood Stabilizer plus SGA | 27 | 27 |  | 54
    Double-Blind Phase: Escitalopram plus SGA | 4 | 4 |  | 8
    Open-Label Phase: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label Phase: Bupropion XL plus Mood Stabilizer |  |  | 35 | 35
    Open-Label Phase: Bupropion XL plus Mood Stabilizer plus SGA |  |  | 33 | 33
    Open-Label Phase: Bupropion XL plus SGA |  |  | 7 | 7
    Open-Label Phase: Escitalopram plus Mood Stabilizer |  |  | 53 | 53
    Open-Label Phase: Escitalopram plus Mood Stabilizer plus SGA |  |  | 64 | 64
    Open-Label Phase: Escitalopram plus SGA |  |  | 14 | 14
Region of Enrollment, Customized [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Data are being reported separately for the Open-label and Double-Blind arms.
  Participants
    Double-Blind Phase: number analyzed (Participants) | 87 | 90 | 0 | 177
    Double-Blind Phase: Canada | 10 | 12 | 0 | 22
    Double-Blind Phase: India | 76 | 76 | 0 | 152
    Double-Blind Phase: South Korea | 1 | 2 | 0 | 3
    Open-Label Phase: number analyzed (Participants) | 0 | 0 | 206 | 206
    Open-Label Phase: Canada | 0 | 0 | 29 | 29
    Open-Label Phase: India | 0 | 0 | 168 | 168
    Open-Label Phase: South Korea | 0 | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Phase: Number of Participants With an Occurrence of Any Mood Episode (Manic, Hypo-manic, Depressive) During the 52 Week Study Period.
Description: The primary outcome, assessed in a time-to-event analysis, was any mood episode, defined as any of the following: a Young Mania Rating Scale (YMRS) score of at least 16 (mild mania), a Montgomery-Åsberg Depression Rating Scale (MADRS) score of at least 20 (moderate depression), a Clinical Global Impressions Scale, Bipolar Version, Severity (CGI-S-BD) score of at least 4 for mania or depression (moderately ill), hospitalization for mood symptoms, necessity of additional pharmacotherapy for emerging mood symptoms, a MADRS suicide item score of at least 4 (scores range from 0 to 6, with higher scores indicating greater suicide risk), or a suicide attempt or suicide death.
  Young Mania Rating Scale:Scores range from 0 to 60,lower scores reflect better clinical outcomes. Montgomery-Åsberg Depression Rating Scale: Scores range from 0 to 60, lower scores reflect better clinical outcomes.
  Clinical Global Impression scale: Scores range from 3 to 42, higher scores reflect worsening status.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 8 Week Arm | 52 Week Arm
Number analyzed (Participants) | 87 | 90
Participants | 40 | 28
Statistical Analysis 1: Comparison: 8 Week Arm vs 52 Week Arm; Test type: Superiority; p = 0.12, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.43 to 1.10] — The hazard ratio for time to any mood episode in the 52-week group relative to the 8-week group was 0.68 (95% confidence interval [CI], 0.43 to 1.10; P = 0.12 by log-rank test)

2. Secondary Outcome: Double-Blind Phase: Number of Participants Who Had an Episode of Mania/Hypomania, Depression or Mixed During the 52 Week Study Period.
Description: Time to a depressive episode, a manic or hypomanic episode, discontinuation from the trial for any clinical reason (e.g., occurrence of a mood event, withdrawal of informed consent, or adverse event), any mood episode or subsyndromal symptoms, time spent in these episodes, and scores on the CGI-BD, YMRS, and MADRS clinical rating scales.
  Young Mania Rating Scale:Scores range from 0 to 60,lower scores reflect better clinical outcomes. Montgomery-Åsberg Depression Rating Scale: Scores range from 0 to 60, lower scores reflect better clinical outcomes.
  Clinical Global Impression scale: Scores range from 3 to 42, higher scores reflect worsening status.
Time Frame: 52 weeks
Population: Of the total 178 patients who underwent randomization, 1 had missing data for baseline and post baseline visits and was excluded from the analysis. Thus, the primary analysis included 177 patients, of whom 90 were assigned to the 52-week group and 87 to the 8-week group.
Measure: Count of Participants; unit: Participants
Groups:
- 8 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s) and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 1 patients randomized to the "8 week arm" will discontinue antidepressant treatment after 8 weeks, as recommended in current clinical practice guidelines. The antidepressant will be tapered in a double-blind manner beginning at 6 weeks, and will be substituted with placebo by 8 weeks.
  Escitalopram 10 - 30 mg Wellbutrin XL 150 - 450 mg
- 52 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s) and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 2 patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.
  Escitalopram 10 - 30 mg Wellbutrin XL 150 - 450 mg
Arm/Group | 8 Week Arm | 52 Week Arm
Number analyzed (Participants) | 87 | 90
Participants
  Manic or hypomanic events | 5 | 11
  Depressive events | 35 | 15
  Mixed episode | 0 | 2
  Subsyndromal depressive symptoms | 8 | 8
  Subsyndromal manic symptoms | 0 | 0
Statistical Analysis 1: Comparison: 8 Week Arm vs 52 Week Arm; Manic or Hypomanic events; Test type: Superiority; Hazard Ratio (HR) = 2.28, 95% CI 2-sided [.86 to 6.08]
Statistical Analysis 2: Comparison: 8 Week Arm vs 52 Week Arm; Depressive Events; Test type: Superiority; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.25 to 0.75]

ADVERSE EVENTS:
Time Frame: 4- 16 weeks on the open-label phase and up to 1 year for each participant in the double-blind phase.
Description: The open-label phase includes adverse events experienced from the 206 participants analyzed in that phase.
  The double-blind phase includes adverse events experienced from the 177 participants analyzed in that phase.
Groups:
- 8 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s)and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 1 patients randomized to the "8 week arm" will discontinue antidepressant treatment after 8 weeks, as recommended in current clinical practice guidelines. The antidepressant will be tapered in a double-blind manner beginning at 6 weeks, and will be substituted with placebo by 8 weeks.
  Escitalopram 10 - 30 mg or Wellbutrin XL 150 - 450 mg
- 52 Week Arm: During the double-blind phase, all patients will continue treatment with their anti-manic medication(s) and will be randomized to one of two treatment arms for up to 52 weeks:
  Group 2 patients randomized to the "52 week arm" will continue treatment with their antidepressant medication for 52 weeks, or until withdrawal from the study.
  Escitalopram 10 - 30 mg or Wellbutrin XL 150 - 450 mg
Arm/Group | 8 Week Arm | 52 Week Arm | Open-Label Phase (4-16 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/90 | 0/206
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/90 | 1/206
Other Adverse Events (participants affected / at risk) | 59/87 | 57/90 | 87/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 8 Week Arm (N=87) | 52 Week Arm (N=90) | Open-Label Phase (4-16 Weeks) (N=206)
Hospitalization due to discontinuation of treatment, alcohol and drug use (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 8 Week Arm (N=87) | 52 Week Arm (N=90) | Open-Label Phase (4-16 Weeks) (N=206)
Abdominal pain or bloating (Gastrointestinal disorders) | 7 | 10 | 6
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Decreased sex drive (Nervous system disorders) | 14 | 12 | 7
Decreased sleep (Nervous system disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 7 | 2 | 2
Feeling faint (Nervous system disorders) | 1 | 2 | 1
Fatigue or tiredness (Nervous system disorders) | 13 | 18 | 12
Headache (Nervous system disorders) | 2 | 2 | 3
Heartburn (Gastrointestinal disorders) | 13 | 8 | 5
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Increased sex drive (Nervous system disorders) | 0 | 4 | 0
Insomnia (Nervous system disorders) | 11 | 9 | 6
Irritability (Psychiatric disorders) | 2 | 4 | 0
Memory problems (Nervous system disorders) | 7 | 14 | 15
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 4
Palpitations (Psychiatric disorders) | 10 | 8 | 5
Poor concentration (Psychiatric disorders) | 0 | 1 | 0
Sleep disturbance (Nervous system disorders) | 0 | 2 | 0
Tremor (Nervous system disorders) | 4 | 6 | 4
Weight gain ≥7% (Endocrine disorders) | 6 | 13 | 2
Other (General disorders) | 8 | 5 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 3
Mania (Psychiatric disorders) | 0 | 0 | 3
Blurred Vision (Eye disorders) | 0 | 0 | 2
Weight Gain (Investigations) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Recruitment was stopped before the planned sample size was reached owing to the Covid-19 pandemic and expiration of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT00958633/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT00958633/SAP_001.pdf